CLINICAL TRIAL: NCT03301246
Title: Artimes Pro Low Profile 1.00mm and 1.25mm Dilatation Catheters for Pre-Dilatation of Stenosis and Occlusion in Patients With Symptomatic Ischemic Heart Disease
Brief Title: Artimes Pro Low Profile Dilatation Catheters for Pre-Dilatation in Patients With Symptomatic Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eminence Clinical Research, Inc. (Industry)
Collaborators: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BROS-CLIN-2017-01
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Heart Disease, Ischemic; Coronary Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: 45 patients will be treated using the 1.0mm dilatation catheter and 15 patients treated with the 1.25mm dilatation catheter for a total of 60 subjects enrolled and treated. Patients may be consented, enrolled and treated until the sample size is reached, with n=60 completing the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Artimes Pro Low Profile Dilatation Catheter (Experimental): Subjects who require initial pre-dilatation using the study device, and then undergo definitive therapy using additional PTCA catheters and stents, according to standard of care will be enrolled in this study.
  Interventions: Device: Artimes Pro Low Profile Dilatation Catheter

INTERVENTIONS:
Device: Artimes Pro Low Profile Dilatation Catheter — Pre-dilation catheter for the purpose of preparing the vessel to deliver the final therapy.

SUMMARY:
This is a prospective, non-randomized, open label, multi-center study including 60 patients with symptomatic ischemic heart disease with 70%-100% coronary artery stenoses and occlusions enrolled and treated in this investigational device study.

DETAILED DESCRIPTION:
Patients who require initial pre-dilatation using the study device, and then undergo definitive therapy using additional PTCA catheters and stents, according to standard of care will be enrolled in this study.

A maximum of 60 subjects with native coronary artery lesions or occlusions will be treated using the Artimes pro Balloon Dilatation Catheters in a 3:1 ratio using the 1.0mm and 1.25mm dilatation catheters for pre-dilatation and will complete the study within the U.S. This equals 45 patients treated using the 1.0mm dilatation catheter, and 15 patients treated with the 1.25mm dilatation catheter for a total of 60 subjects enrolled and treated.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Willing and able to provide informed consent;
* Willing and able to meet all study requirements;
* Patients with symptomatic ischemic heart disease due to stenotic lesions or occlusions in coronary arteries that are amenable to percutaneous coronary interventions;
* Patients who tolerate DAPT

Exclusion Criteria:

* A known hypersensitivity or contraindication to aspirin, heparin, or bivalirudin, anti-platelet medications, or sensitivity to contrast media, which cannot be adequately pre-medicated;
* LVEF < 30%;
* Evidence of an acute myocardial infarction within 72 hours of the intended index procedure;
* Planned treatment of unprotected left main disease;
* History of cerebral vascular accident (CVA) within 6 months prior to consideration for this study;
* Transient ischemic attack (TIA) within 6 months prior to consideration for this study;
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months prior to consideration for this study;
* History of bleeding diathesis or coagulopathy;
* Refuses blood transfusions;
* Any general contraindication to revascularization procedures;
* Pregnant or lactating;
* In the judgement of the investigator, patient is not a suitable candidate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Procedure Success | Day 1 - Index Procedure
  Delivery of the catheter to and across lesion; inflation and deflation of the catheter; no vessel perforation, dissection or reduction in TIMI flow; and achievement of final TIMI flow grade 3.

SECONDARY OUTCOMES:
Anticipated Adverse Events | Day 1 - Index Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jasvinder Singh, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No